CLINICAL TRIAL: NCT02734719
Title: Increasing Bone Density by Application of Surface Electrical Stimulation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Device is not available.
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Konstantinovic Ljubica, professor, University of Belgrade
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LK-2
Record Dates: First submitted 2016-03-29; First posted 2016-04-12 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Osteoporosis; Electrical Stimulation; Posture
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group treated with Bonestim (Experimental): The experimental group will be treated with the electrical stimulation device Bonestim.
  Interventions: Device: Bonestim

INTERVENTIONS:
Device: Bonestim — Bonestim is the multipad electrical stimulation device.
  Other Names: multipad electrical stimulation of trunk muscles

SUMMARY:
Bonestim system for osteoporosis treatment uses surface electrical stimulation of neuromuscular and skeletal tissue by multipad stimulation electrodes for inducing contractions of the spinal column muscles. The primary aim of this clinical study is to determine if the Bonestim therapy can improve bone density. A secondary aim is to determine whether the applied treatment increases postural stability and facilitation of daily life activities.

Inducing of contractions of the spinal column muscles in this manner could be new treatment options for the patients with reduced mobility and the patients with serious contraindications for drugs.

ELIGIBILITY:
Inclusion Criteria:

* T score at least 1,5 (ideal 2,-2,5)
* Stable bone turn over (lab.analyses.)

Exclusion Criteria:

* fracture,pace maker, malignancy and gastrointestinal problems
* chronic corticosteroid therapy
* spinal surgery in previous year

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
density of bone measured by central Dxa measurement | 6 months

SECONDARY OUTCOMES:
sagittal flexibility measured by Schober measurement | 6 months
daily activities measured by Oswestry disability index | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic for rehabilitation dr Miroslav Zotovic Faculty of Medicine University of Belgrade, Belgrade, Serbia